CLINICAL TRIAL: NCT00184821
Title: Acute Local Ischemic Preconditioning in Patients With Type 1 Diabetes in Vivo
Brief Title: Ischemic Injury and Ischemic Preconditioning in Diabetes
Status: Completed | Type: Observational
Sponsor: Radboud University Medical Center (Other)
Collaborators: Dutch Diabetes Fund (Unknown)
Other Study IDs: QKF03-diab; 2004.11.022
Record Dates: First submitted 2005-09-09; First posted 2005-09-16 (Estimated); Last update posted 2007-04-05 (Estimated); Status verified 2007-04

CONDITIONS: Diabetes Mellitus, Insulin-Dependent; Ischemia-Reperfusion Injury
Keywords: Diabetes; Ischemia; Annexin A5 scintigraphy
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Reperfusion Injury; Diabetes Mellitus; Ischemia | interventions — Ischemic Preconditioning; Diazoxide; Glyburide; Adenosine

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Other
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Ischemic preconditioning
Procedure: Forearm ischemic exercise
Procedure: Annexin A5 scintigraphy
Drug: Diazoxide
Drug: glibenclamide
Drug: adenosine

SUMMARY:
In this proof-of-concept study, forearm vulnerability to ischemic exercise is studied in patients with type 1 diabetes mellitus with and without prior ischemic preconditioning (short period of ischemia that protects against subsequent ischemic exercise). Annexin A5 scintigraphy is used to quantify subtle signs of mild and reversible forearm injury that results from ischemic exercise.

The following hypotheses are tested:

1. Patients with type 1 diabetes are not more vulnerable to ischemic injury as compared with previously studied healthy volunteers.
2. Ischemic preconidtioning is still present in patients with type 1 diabetes. Depending on the validity of hypothesis 2, the effect of short pharmacological interventions are studied on vulnerability to forearm ischemia/reperfusion injury in the absence or presence of local forearm ischemic preconditioning.

DETAILED DESCRIPTION:
All patients will be studied in supine position after an overnight fast, while plasma glucose levels are monitored. In the first 8 patients intravenous insulin is administered as needed, to reach target glucose levels between 5-7 mmol/l. Patients will be subjected to 10 minutes of forearm ischemia (non-dominant arm), combined with handgripping at 50% of maximal force until exhaustion. Upon reperfusion, Tc-99m-HYNIC-Annexin A5 will be injected intravenously. Targeting of annexin A5 to thenar muscle and forearm flexor muscle will be quantified as the percentage difference in radioactivity between experimental and control side. This procedure will be performed twice (randomized cross-over design), with at least 2 week interval, either with or without 10 minutes ischemia followed by 10 minutes of reperfusion prior to ischemic exercise.

Depending on the results of this study, substudies will be performed to study the effect of diazoxide (K-ATP channel opener, may mimic ischemic preconditioning), glibenclamide (K-ATP channel blocker, may inhibit ischemic preconditioning) or adenosine (infusion into brachial artery of non-dominant arm as a substitute for ischemic preconditioning).

ELIGIBILITY:
Inclusion Criteria:

* type 1 diabetes mellitus
* age 18-50 years

Exclusion Criteria:

* hypertension (systolic blood pressure > 140 mmHg and/or diastolic blood pressure > 90 mmHg
* cardiovascular disease (coronary artery insufficiency,CVA/TIA, peripheral artery disease
* HbA1c > 9%
* Body Mass Index < 25 kg/m2
* Unable to stop co-medication (other than insulin) for 1 week
* Previous exposure to radiation (diagnostic or therapeutic) in the past year

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20
Dates: Start 2004-06; Study Completion 2005-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard Engbersen, MD, Study Chair — Radboud University Nijmegen Medical Centre; department of Pharmacology-Toxicology; Gerard Rongen, MD, PhD, Study Chair — Radboud University Nijmegen Medical Centre; Department of Pharmacology-Toxicology; Wim Oyen, MD, PhD, Study Chair — Radboud University Nijmegen Medical Centre; Department of Nuclear Medicine; Marc Mol, MD, PhD, Study Chair — Canisius Wilhelmina Ziekenhuis Nijmegen; Department of Internal Medicine; Paul Smits, MD, PhD, Principal Investigator — Radboud University Nijmegen Medical Centre; Department of Pharmacology-Toxicology; B. Bravenboer, MD, PhD, Study Chair — Catharina Hospital Eindhoven, Dept. of Internal Medicine
Locations (1):
- Clinical Research Centre Nijmegen; Radboud University Nijmegen Medical Centre, Nijmegen, Gelderland, Netherlands

REFERENCES:
- [Derived] Engbersen R, Riksen NP, Mol MJ, Bravenboer B, Boerman OC, Meijer P, Oyen WJ, Tack C, Rongen GA, Smits P. Improved resistance to ischemia and reperfusion, but impaired protection by ischemic preconditioning in patients with type 1 diabetes mellitus: a pilot study. Cardiovasc Diabetol. 2012 Oct 10;11:124. doi: 10.1186/1475-2840-11-124. PMID 23051145